CLINICAL TRIAL: NCT05594095
Title: Precision Platform Study of HR+/ HER2-advanced Breast Cancer Based on SNF Typing (A Prospective, Open-label, Multi-center, Phase II Platform Study)
Brief Title: SNF Platform Study of HR+/ HER2-advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); First Hospital of China Medical University (Other); Sun Yat-sen University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Chongqing University Cancer Hospital (Other); Northern Jiangsu People's Hospital (Other); Fujian Medical University Union Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Shanghai First Maternity and Infant Hospital (Other); Shanghai 6th People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Nanchang People's Hospital (Unknown); Liaoning Cancer Hospital & Institute (Other); The Affiliated Hospital of Nantong University (Unknown); The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCTOP-L-M05
Record Dates: First submitted 2022-10-13; First posted 2022-10-26 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasm; Breast Cancer; Hormone Receptor Positive Tumor; HER2-negative Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; famitinib; fluzoparib; dalpiciclib; Everolimus; Aromatase Inhibitors; Fulvestrant; Goserelin; Sorafenib; apatinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (26):
- SNF1 1A: PIK3CA mutation (Experimental): PIK3CA inhibitors +Aromatase inhibitors(Letrozole/Anastrozole/Exemestane, po, qd, specific dose (letrozole 2.5mg/ day; Anastrozole 1mg/ day, Exemestane 25mg/ day);Or fulvestrant, 500mg ,im, qm, followed by 500mg im 2 weeks after the first dose; Premenopausal: Goserelin 3.6mg IM every 4 weeks.
  Interventions: Drug: PIK3CA inhibitor; Drug: Aromatase Inhibitors or Fulvestrant; Drug: Goserelin
- SNF1 1B: AKT pathway mutation (Experimental): AKT pathway inhibitors +Aromatase inhibitors(Letrozole/Anastrozole/Exemestane, po, qd, specific dose (letrozole 2.5mg/ day; Anastrozole 1mg/ day, Exemestane 25mg/ day);Or fulvestrant, 500mg ,im, qm, followed by 500mg im 2 weeks after the first dose; Premenopausal: Goserelin 3.6mg IM every 4 weeks.
  Interventions: Drug: AKT inhibitor; Drug: Aromatase Inhibitors or Fulvestrant; Drug: Goserelin
- SNF1 1C: without above mutation (Experimental): Everolimus 10mg po qd+Aromatase inhibitors(Letrozole/Anastrozole/Exemestane, po, qd, specific dose (letrozole 2.5mg/ day; Anastrozole 1mg/ day, Exemestane 25mg/ day);Or fulvestrant, 500mg ,im, qm, followed by 500mg im 2 weeks after the first dose; Premenopausal: Goserelin 3.6mg IM every 4 weeks.
  Interventions: Drug: Everolimus; Drug: Aromatase Inhibitors or Fulvestrant; Drug: Goserelin
- SNF2 2A (Experimental): Treatment of physician' choice+Pd-1 mab (Carrelizumab 200mg Q2W)+Famitinib 15mg po qd for 4 weeks as a cycle
  Interventions: Drug: Carrelizumab; Drug: Famitinib; Drug: TPC
- SNF3 3A: Stratification of BRCA/PALB2 expression (Experimental): Fluzoparib SHR3162 100mg po qd+Dalpiciclib 125mg po qd for 4 weeks as a cycle
  Interventions: Drug: Fluzoparib; Drug: Dalpiciclib
- SNF4 4A: HER2 low (Experimental): SHR-A1811
  Interventions: Drug: SHR-A1811
- The control arm (Active Comparator): Treatment of Physicians' Choice (albumin-paclitaxel, capecitabine, vinorelbine, and irbribulin)
  Interventions: Drug: TPC
- SNF3 3B: (Experimental): Fluzoparib SHR3162 100 mg qd+Treatment of physician' choice
  Interventions: Drug: Fluzoparib; Drug: TPC
- SNF4 4B: (Experimental): Apatinib 250mg qd+Treatment of physician' choice
  Interventions: Drug: TPC; Drug: Apatinib
- SNF1 1D: without above mutation (Experimental): Everolimus 10mg po qd+Treatment of physician' choice
  Interventions: Drug: Everolimus; Drug: TPC
- SNF1 1E: HER2 LOW (Experimental): Everolimus 10mg po qd+SHR-A1811
  Interventions: Drug: SHR-A1811; Drug: Everolimus
- SNF1 1F: HER2 zero (Experimental): Everolimus 10mg po qd+SHR-A1921
  Interventions: Drug: Everolimus; Drug: SHR-A1921
- SNF2 2B: HER2 zero (Experimental): SHR-A1921+Pd-1 mab (Carrelizumab 200mg Q2W)+bevacizumab 7.5mg po ivgt t for 3 weeks as a cycle
  Interventions: Drug: Carrelizumab; Drug: SHR-A1921; Drug: bevacizumab
- SNF2 2C: (Experimental): HER3 -ADC+Pd-1 mab (Carrelizumab 200mg Q2W)+Famitinib for 3 weeks as a cycle
  Interventions: Drug: Carrelizumab; Drug: Famitinib; Drug: SHR-A2009
- SNF2 2D: (Experimental): Nectin4-ADC+Pd-1 mab (Carrelizumab 200mg Q2W)+Famitinib for 3 weeks as a cycle
  Interventions: Drug: Carrelizumab; Drug: Famitinib; Drug: SHR-A2102
- SNF2 2E: HER2 low (Experimental): SHR-A1811+Pd-1 mab (Carrelizumab 200mg Q2W)+Famitinib for 3 weeks as a cycle
  Interventions: Drug: Carrelizumab; Drug: Famitinib; Drug: SHR-A1811
- SNF3 3C: (Experimental): CDK4i（SHR-6209 PR2D+PARP1i（SHR-1167 PR2D）
  Interventions: Drug: SHR-1167; Drug: SHR-6209
- SNF3 3D: (Experimental): PARP1i（SHR-1167 PR2D)+Famitinib 5mg po qd for 4 weeks as a cycle
  Interventions: Drug: Famitinib; Drug: SHR-1167
- SNF3 3E: HER2 low (Experimental): PARP1i（SHR-1167 PR2D)+SHR-A1811 for 3 weeks as a cycle
  Interventions: Drug: SHR-A1811; Drug: SHR-1167
- SNF3 3F: HER2 zero (Experimental): PARP1i（SHR-1167 PR2D)+SHR-A1921 for 3 weeks as a cycle
  Interventions: Drug: SHR-A1921; Drug: SHR-1167
- SNF4 4C (Experimental): Famitinib 20mg po qd
  Interventions: Drug: Famitinib
- SNF4 4D (Experimental): Sorafenib 0.4g bid
  Interventions: Drug: Sorafenib
- SNF4 4E (Experimental): Apatinib 500mg qd
  Interventions: Drug: Apatinib
- SNF4 4F: HER2 low (Experimental): Famitinib+SHR-A1811 for 3 weeks as a cycle
  Interventions: Drug: Famitinib; Drug: SHR-A1811
- SNF4 4G (Experimental): Famitinib+HER3-ADC for 3 weeks as a cycle
  Interventions: Drug: Famitinib; Drug: SHR-A2009
- SNF4 4H (Experimental): Famitinib+Nectin4-ADC for 3 weeks as a cycle
  Interventions: Drug: Famitinib; Drug: SHR-A2102

INTERVENTIONS:
Drug: PIK3CA inhibitor — PIK3CA inhibitor
  Arms: SNF1 1A: PIK3CA mutation
Drug: AKT inhibitor — AKT inhibitor
  Arms: SNF1 1B: AKT pathway mutation
Drug: Carrelizumab — Pd-1 mab
  Other Names: SHR1210
  Arms: SNF2 2A; SNF2 2B: HER2 zero; SNF2 2C:; SNF2 2D:; SNF2 2E: HER2 low
Drug: Famitinib — VEGFR inhibitor
  Arms: SNF2 2A; SNF2 2C:; SNF2 2D:; SNF2 2E: HER2 low; SNF3 3D:; SNF4 4C; SNF4 4F: HER2 low; SNF4 4G; SNF4 4H
Drug: Fluzoparib — PARP inhibitor
  Other Names: SHR3162
  Arms: SNF3 3A: Stratification of BRCA/PALB2 expression; SNF3 3B:
Drug: Dalpiciclib — CDK4/6 inhibitor
  Other Names: SHR6390
  Arms: SNF3 3A: Stratification of BRCA/PALB2 expression
Drug: SHR-A1811 — HER2 ADC
  Arms: SNF1 1E: HER2 LOW; SNF2 2E: HER2 low; SNF3 3E: HER2 low; SNF4 4A: HER2 low; SNF4 4F: HER2 low
Drug: Everolimus — mTOR inhibior
  Arms: SNF1 1C: without above mutation; SNF1 1D: without above mutation; SNF1 1E: HER2 LOW; SNF1 1F: HER2 zero
Drug: Aromatase Inhibitors or Fulvestrant — Letrozole/Anastrozole/Exemestane or Fulvestrant
  Arms: SNF1 1A: PIK3CA mutation; SNF1 1B: AKT pathway mutation; SNF1 1C: without above mutation
Drug: Goserelin — For premenopause
  Arms: SNF1 1A: PIK3CA mutation; SNF1 1B: AKT pathway mutation; SNF1 1C: without above mutation
Drug: TPC — Treatment of Physicians' Choice (albumin-paclitaxel, capecitabine, vinorelbine, and irbribulin)
  Arms: SNF1 1D: without above mutation; SNF2 2A; SNF3 3B:; SNF4 4B:; The control arm
Drug: Sorafenib — RTK Inhibitor
  Arms: SNF4 4D
Drug: Apatinib — Apatinib 250mg po qd
  Arms: SNF4 4B:; SNF4 4E
Drug: SHR-A1921 — TROP2 ADC
  Arms: SNF1 1F: HER2 zero; SNF2 2B: HER2 zero; SNF3 3F: HER2 zero
Drug: SHR-A2102 — NECTIN4 ADC
  Arms: SNF2 2D:; SNF4 4H
Drug: SHR-A2009 — HER3 ADC
  Arms: SNF2 2C:; SNF4 4G
Drug: SHR-1167 — PARP1i
  Arms: SNF3 3C:; SNF3 3D:; SNF3 3E: HER2 low; SNF3 3F: HER2 zero
Drug: SHR-6209 — CDK4i
  Arms: SNF3 3C:
Drug: bevacizumab — bevacizumab
  Arms: SNF2 2B: HER2 zero

SUMMARY:
The purpose of this study is to establish a prospective, multi-center platform research based on clinical subtypes to explore precision therapy in patients hormone-receptor-positive HER2-negative advanced breast cancer who had previously used CDK4/6 inhibitors.

DETAILED DESCRIPTION:
Participants in this study were hormone-receptor-positive HER2-negative patients with advanced breast cancer who had previously used CDK4/6 inhibitors. Hormone receptor positive HER2 negative was defined as ER positive (IHC ER positive percentage > 10% or PR positive (IHC PR positive percentage > 10%) and HER2 negative (IHC-/+; Or IHC++ but FISH/CISH-).

The Department of Pathology and the Key Laboratory of Breast Cancer of Fudan University Shanghai Cancer Center conducted digital pathological typing of the biopsy pathology of metastatic lesions of all participants . If the pathology of metastatic lesions could not be obtained, the digital pathological typing was performed according to the pathology of primary lesions. According to the digital pathological types of biopsy tissue and peripheral blood ctDNA, the patients were divided into four precise subtypes: SNF1, SNF2, SNF3, and SNF4. At the same time, the negative control group was randomly set by subtype stratification at 2:1. In different SNF types, patients were divided into 7 subcohorts according to the genetic PANEL results.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥18 years;
2. HR+/HER2- invasive breast cancer confirmed by histology (specific definition: ER >10% positive tumor cells by immunohistochemistry is defined as ER positive, PR >10% positive tumor cells is defined as PR positive, ER and/or PR positive is defined as HR positive; HER2 0-1+ or HER2 + but negative by FISH without amplification was defined as HER2 negative);
3. Locally advanced breast cancer (unable to undergo radical local treatment) or recurrent metastatic breast cancer;
4. HR+/HER2- advanced breast cancer patients who had previously received CDK4/6 inhibitor therapy;
5. At least one measurable lesion according to RECIST 1.1 (conventional CT scan ≥20 mm, spiral CT scan ≥10 mm, measurable lesion has not received radiotherapy);
6. The functions of the main organs are basically normal and meet the following conditions:

   I. Blood routine examination criteria shall meet: HB ≥90 g/L (no blood transfusion within 14 days); The ANC acuity 1.5 x 109 / L; PLT acuity 75 x 109 / L; Ii. Biochemical tests should meet the following criteria: TBIL ≤1.5×ULN (upper limit of normal value); ALT and AST ≤3×ULN; If liver metastases were present, ALT and AST≤ 5×ULN; Serum Cr ≤1×ULN, endogenous creatinine clearance > 50 ml/min (Cockcroft-Gault formula);
7. They have not received radiotherapy, molecular targeted therapy, or surgery within 3 weeks before the start of the study, and have recovered from the acute toxicity of previous treatment (if surgery was performed, the wound has healed completely); No peripheral neuropathy or grade I peripheral neurotoxicity;
8. ECOG score ≤2, and life expectancy ≥3 months;
9. Fertile female subjects were required to use a medically approved contraceptive method during the study treatment period and for at least 3 months after the last use of the study drug;
10. Subjects volunteered to join the study, signed informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Radiotherapy (except for palliative causes), chemotherapy, and immunotherapy were used in the first 3 weeks of treatment, except bisphosphonate (which can be used for bone metastasis);
2. Uncontrolled central nervous system metastases (indicating symptomatic or symptomatic treatment with glucocorticoids or mannitol);
3. A history of clinically important or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction, or ventricular arrhythmia within the last 6 months;
4. Persistent grade 1 or higher adverse reactions caused by previous treatments. The exception to this is hair loss or something the researchers don't think should be ruled out. Such cases should be clearly documented in the investigator's notes;
5. Underwent major surgery (except minor outpatient procedures, such as placement of vascular access) within 3 weeks of the first course of trial treatment;
6. Pregnant or lactating patients; Malignancy (except basal cell carcinoma of the skin, which has been cured, and carcinoma in situ of the cervix) in the past 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 3 years)
  The proportion of participants whose best outcome is complete remission or partial remission (according to RECIST1.1)

SECONDARY OUTCOMES:
Clinical Benefit Rate (CBR) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 3 years
  the percentage of subjects with CR+PR+SD and last more than 24 weeks in all of the subjects
Progression Free Survival (PFS) | Randomization until the first occurrence of disease progression or death from any cause, which ever occurs first, through the end of study (approximately 3 years)]
  time to progressive disease (according to RECIST1.1)
Overall Survival (OS) | Randomization to death from any cause, through the end of study (approximately 3 years)
  time to death due to any cause
CTCAE scale (V5.0) | up to One Year during follow-up
  To evaluate the rate of adverse effects of patient by the standard CTCAE scale (V5.0)
Exploration of translational research markers | up to One Year during follow-up
  The collected subjects' tumor tissues, paracancerous tissues, blood, and fecal samples will be used for discovering exploratory biomarkers. The relationships between discovered biomarkers and subjects' disease status and treatment responses will also be investigated.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided